CLINICAL TRIAL: NCT05753111
Title: Effect of Palmitoylethanolamide on Muscle Recovery Following a Single Bout of Resistance Exercise
Brief Title: Effect of PEA on Muscle Recovery Following Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, sebastiaan dalle, Postdoctoral researcher, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S67315
Record Dates: First submitted 2023-01-19; First posted 2023-03-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Muscle Recovery; Muscle Soreness
Keywords: PEA; Skeletal muscle
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, crossover trial design
Who Masked: Participant, Investigator
Masking Description: Blinding: To avoid bias, treatment arms will be blinded to Investigators/Trial staff/participants, as follows: the supplement will be manufactured, packaged and labelled in such a way that the visual appearance, nor the smell and/or touch of the supplement can be distinguished from the placebo. Supplements are delivered to the participants by a member of the research group that is not involved in any of the experimental procedures or analyses. Furthermore, to maintain the blind, the supplement and placebo will follow the same administration route and process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants receive placebo supplements on two separate occasions in a randomized order. The placebo supplements contain 350 mg of maltodextrine. Placebo supplements are packaged in non-see-through hard capsules to assure that there are no differences in appearance or taste. Participants are instructed to ingest their supplement twice a day (in the morning and one hour before bedtime) for 6 consecutive days starting after collection of baseline measures.
  Interventions: Dietary Supplement: PLACEBO
- Palmitoylethanolamide (PEA) supplementation (Experimental): Participants receive PEA supplements on two separate occasions in a randomized order. The PEA supplements contain 350 mg of Levagen+ (315 mg of PEA and 35 mg of excipients). Levagen+ consists for 90% of palmitoylethanolamide and for 10% of a mixture of coconut oil (fractionated), polyglycerol polyricinoleate, citrus oil, olive oil, lecithin, dl-alpha tocopheryl acetate, and silicon dioxide to improve the bioavailability of PEA. Both PEA supplements are packaged in non-see-through hard capsules to assure that there are no differences in appearance or taste. Participants are instructed to ingest their supplement twice a day (in the morning and one hour before bedtime) for 6 consecutive days starting after collection of baseline measures.
  Interventions: Dietary Supplement: PEA

INTERVENTIONS:
Dietary Supplement: PEA — PEA supplementation
  Other Names: Levagen+
  Arms: Palmitoylethanolamide (PEA) supplementation
Dietary Supplement: PLACEBO — Maltodextrin supplementation
  Arms: Placebo

SUMMARY:
This study evaluates the effects of short term palmitoylethanolamide (PEA) supplementation on functional responses (i.e. muscle soreness and performance parameters) to strenuous eccentric exercise, and investigateq the systemic and muscle molecular mechanisms through which PEA impacts on these functional responses.

DETAILED DESCRIPTION:
Study design The protocol entails a double-blind, placebo-controlled, crossover trial design in which non-elite male athletes (training load >5h/wk, n=14) are enrolled. Participants undergo 2 experimental sessions in which they receive PEA or placebo in a randomized order. The two sessions are separated by a 3-week wash out period to allow a full recovery from the eccentric exercise bout. The scientific rationale to use a within-subjects design is based on the assumption of reduced data variability and increased statistical power compared to a between-subjects design. Additionally, a double-blind placebo controlled trial is used to prevent treatment bias and placebo effects.

Participants are randomly allocated to receive PEA or appearance-matched placebo supplements twice a day for a total of 6 days. Three days before the start of supplementation (D-3), baseline measurements are collected during which participants report to the laboratory in a fasted and rested state and mark their perceived muscle soreness on a visual analogue scale (VAS). Next, blood samples and muscle biopsies are collected, after which maximal isometric, eccentric and concentric voluntary contractions and jump height (Counter Movement Jump and Squat Jump) are assessed. Furthermore, participants complete the Pittsburgh Sleep Quality Index (PSQI) to evaluate sleep quality and quantity of the previous month. Three days after the collection of baseline measurements (D0), participants return to the laboratory in a rested and fasted state. After collection of a fasted blood sample, they receive their first supplement with a light standardized breakfast (~500 kcal, 60% carbohydrates, 20% protein, 20% fat). Afterwards, they rate their perceived muscle soreness and fill in the St. Mary's Hospital questionnaire (to evaluate their sleep quality and quantity from the previous night). One hour after supplement intake, participants perform a unilateral eccentric exercise (EE) bout consisting of 24 sets of 10 eccentric contractions of the knee extensors. Measurements of maximal voluntary contractions and jump height are repeated 24, 48, 72 and 120h following EE. Additionally, blood samples are collected 24, 48, 72, 96 and 120h following EE, and muscle biopsies are collected 48h following EE. Furthermore, participants rate their perceived muscle soreness, complete a food diary and fill in the St. Mary's Hospital questionnaire (daily), for the entire duration of the experimental protocol.

Screening Volunteers are screened to assess their eligibility to participate in the study based on in- and exclusion criteria . During the screening, body mass is measured using a digital balance with an accuracy of 0.1 kg and body height is measured with an accuracy of 1 cm. Furthermore, a medical questionnaire is obtained to assess participants' general health. When volunteers are deemed eligible according to the screening results and the in- and exclusion criteria, they are included in the study.

Familiarization To prevent any learning effect during the intervention trial, all participants are familiarized with the test equipment at least one week before the start of the trial. Participants are invited to perform 3 submaximal isometric, eccentric and concentric voluntary contractions and 3 counter movement jumps and squat jumps as described in detail below (see paragraph 76.3 on page 12). Participants are instructed about the proper technique of the movements and are supervised by a staff member at all times. During the familiarization, individual settings on the isokinetic dynamometer are determined and will be used in all subsequent measurements. Additionally, participants are instructed on how to complete their food diaries.

Randomization: Participants are randomly allocated to one of the supplemental groups (PEA orplacebo) during the first session. After a wash out period of 3 weeks participants are crossed over to the other supplement group. Randomization is performed by a researcher within our lab who is not involved in any of the experimental procedures. As such, the participants as well as the researchers performing the measurements are unaware of the order in which participants receive the different supplements. The randomization sequence will be generated by a member of the research group that is not involved in the current study using an online tool (RANDOM.ORG - Integer Set Generator). Identity concealment codes are used in the randomization list which is in the safe custody of the same member of the research group that is not involved in the current study.

Blinding: To avoid bias, treatment arms will be blinded to Investigators/Trial staff/participants, as follows: the supplement will be manufactured, packaged and labelled in such a way that the visual appearance, nor the smell and/or touch of the supplement can be distinguished from the placebo. Supplements are delivered to the participants by a member of the research group that is not involved in any of the experimental procedures or analyses. Furthermore, to maintain the blind, the supplement and placebo will follow the same administration route and process.

Unblinding: After all participants have completed the Trial and all wet-lab analyses are completed, the database will be locked and the collected Trial data will be unblinded to allow statistical analysis of the Trial data. The PI will provide the designated researchers with the unblinded treatment information for all participants after completing the data analysis.

In case of an emergency in a blinded Trial, the Investigator has the sole responsibility for determining if premature unblinding of a participant's treatment assignment is warranted. Participant safety must always be the first consideration in making such a determination. The date and reason for unblinding must be recorded, as applicable.

Muscle damaging eccentric exercise (EE) protocol Participants perform a 5-minute warm up on the cycle ergometer at 100W. Afterwards, they take place on the isokinetic dynamometer where their upper body is strapped to the chair to stabilize their trunk and their right leg is strapped to the lever arm. The EE protocol consists of 24 sets of 10 isokinetic unilateral eccentric contractions of the knee extensors at an angular velocity of -30⁰/s and a range of motion from 180⁰ to 60⁰ (where 180⁰ refers to full extension). In between sets, 60 seconds of rest is provided. Participants are verbally encouraged to maximally resist the downward rotation of the lever arm during the eccentric phase of the movement. No resistance is applied during the concentric phase of the movement. This eccentric exercise protocol showed to effectively induce muscle damage as indicated in previous studies.

Supplements Participants receive PEA and placebo supplements on two separate occasions in a randomized order. The PEA supplements contain 350 mg of Levagen+ (315 mg of PEA and 35 mg of excipients) and the placebo supplements contain 350 mg of maltodextrine. Levagen+ consists for 90% of palmitoylethanolamide and for 10% of a mixture of coconut oil (fractionated), polyglycerol polyricinoleate, citrus oil, olive oil, lecithin, dl-alpha tocopheryl acetate, and silicon dioxide to improve the bioavailability of PEA. Both PEA and placebo supplements are packaged in non-see-through hard capsules to assure that there are no differences in appearance or taste. Participants are instructed to ingest their supplement twice a day (in the morning and one hour before bedtime) for 6 consecutive days starting after collection of baseline measures.

Physical activity and Dietary control The participants are asked to maintain their habitual activity patterns (e.g. biking to class). However, they are instructed not to perform any moderate to strenuous exercise during and 72h before the start of the experimental session. Furthermore, no exercise of any kind is allowed 24h before the collection of muscle biopsies.

Participants receive a standardized meal (1200 kcal; 180 g CHO, 33 g fat, 45 g protein) on the evening before EE as well as on the evening before muscle biopsy collection. On testing days, when participants have to report to the lab in a fasted state, a breakfast (500 kcal) is provided upon completion of all measurements. The same breakfast is provided 1 hour before the start of EE. Furthermore, participants complete a food diary daily, starting after baseline measurements, in order to check for possible dietary variation between conditions. Dietary analyses are performed using a web-platform for dietary recording and analysis of macronutrient and micronutrient composition (https://mijn.voedingscentrum.nl/nl/eetmeter/). Participants are not allowed to consume alcoholic or caffeinated beverages during the experimental sessions.

Blood samples Blood (2x10 mL) is sampled from an arm vein (Venoject system), and plasma or serum is immediately separated by centrifuging. Plasma and serum samples are distributed in different 1 mL aliquots and stored at -20°C until usage for biochemical assays at a later date. Blood samples are collected at baseline, immediately before EE and 24, 48, 72, 96 and 120h following EE in a fasted state.

Plasma samples are analysed by appropriate specific Enzyme-Linked Immunosorbent Assay (ELISA) for CK (marker for muscle damage), IL-6 and TNFalpha (both markers of systemic inflammation). PEA concentrations are assessed by high-performance liquid chromatography with tandem mass spectrometry. Additional assays on blood samples may be performed if judged relevant after the primary analyses have been performed. After all analyses have been performed, any residual sample is stored for an additional 3 years period before being permanently destroyed.

Muscle biopsies Muscle biopsies are collected at baseline and 48h following EE from the dominant leg in a fasted state. Hence, a total of 4 biopsies per subject are taken throughout the study. Biopsies are taken by an experienced physician (Dr. Ruud Van Thienen) from the m. vastus lateralis of the trained leg using a Bergström needle with a 5 mm diameter as previously described (29). In short, a small incision (~5mm) is made through the skin and underlying fascia under local anaesthesia (Lidocaïne, 1ml) to facilitate smooth penetration of the needle into the muscle belly. Once the needle is placed within the muscle belly, a tube and syringe are attached to the upper extremity of the needle which is used to create a vacuum by which the muscle is drawn into the needle. At this point, a smooth twisting downward movement of the inner part of the needle cuts through the tissue to obtain the muscle sample. After cutting of the tissue (~150-300 mg of muscle) the samples are freed from any visual blood and connective tissue before being frozen in liquid nitrogen. The incision that was made through the skin will be closed using adhesive strips (steristrips) and bandaged with a waterproof plaster. Participants will wear the plaster for 5 days before they are allowed to take it off. During these 5 days participants are allowed to take a shower but they will be instructed not to immerse or plunge the plaster (i.e. taking a bad or swim). Participants will be warned about the fact that the muscle biopsy procedure leaves a small scar of ~5mm that most likely will be invisible after one or two years. Furthermore, the local anaesthesia assures that there is no pain sensation during the procedure, but mechanical sensors in the muscles remain sensitive. As such, participants may experience the feeling of pressure but not pain. After the procedure the muscle may feel stiff for a day or two.

Muscle biopsies are biochemically analysed within our lab (Exercise Physiology research lab, KU Leuven) for parameters of muscle inflammation, stress, regeneration and anabolism.

Maximal voluntary contraction (MVC) of the knee extensors The isometric, eccentric and concentric knee extensor torque of the trained leg are measured using an isokinetic dynamometer (cfr. (28)) at baseline and 24, 48, 72 and 120h following EE. In short, participants are seated with their upper body strapped to the chair to stabilize the trunk and their trained leg strapped to the lever arm. For maximal isometric voluntary contraction peak, the knee joint is placed at an angle of 90⁰. Participants are instructed to maximally contract their knee extensors and hold it for 3 seconds. Maximal eccentric and concentric voluntary contraction are measured at an angular velocity of 30⁰/s and a range of motion between 180-60⁰ (where 180⁰ refers to full extension). Each movement is performed three times with 60 seconds of rest between attempts. The maximal peak torque value obtained between attempts is used for analysis.

Counter movement jump Participants perform a counter movement jump (CMJ) on a force platform (SMARTJUMP, Fusion sport, Nottingham, UK) at baseline and 24, 48, 72 and 120h following EE. Participants are asked to take an upright position (knee angle of 180⁰) with their feet on hip width before they initiate a downward movement to squat position (knee angle of 90⁰) after which they jump vertically for maximum height. Participants are instructed to place their hands on their hips and to keep their body erect throughout the jump. CMJ is performed three times with 60 seconds of rest between attempts. The highest jump recorded is used for analysis.

Squat jump Participants perform a squat jump (SJ) on a force platform at baseline and 24, 48, 72 and 120h following EE. Participants are asked to start at a squat position (knee angle of 90⁰) and hold this for 3 seconds before they jump vertically for maximum height. Participants are instructed to place their hands on their hips and to keep their body erect throughout the jump. SJ is performed three times with 60 seconds rest between attempts. The highest jump recorded is used for analysis.

Muscle soreness Muscle soreness of the trained leg is assessed at baseline, immediately before EE and 24, 48, 72, 96 and 120h following EE using a visual analogue scale (VAS). Participants are asked to hold a squat position for 3 seconds with their hands on their hips and to mark their perceived muscle soreness on a scale that is represented by a 100mm line of which the far-left represents 'no pain' while the far-right represents 'extreme pain'.

Sleep quality and quantity At baseline, participants' habitual sleep hygiene is evaluated using the Pittsburgh Sleep Quality Index . In addition, participants complete the St. Mary's Hospital questionnaire daily to evaluate their sleep quality and quantity from the previous night, starting on the night before baseline measurements. The St. Mary's Hospital questionnaire showed to be a reliable tool for assessing the previous night's sleep of a subject.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 35 years old
* Non-elite athletes (training load > 5h/wk)
* Good health status confirmed by a medical screening
* Body Mass Index (BMI) between 18 and 25 kg/m2
* Masters the Dutch language

Exclusion Criteria:

* Participant has a history of smoking
* Concomitant participation in another interventional Trial (e.g. with an investigational medicinal product, medical device or experimental surgical technique)
* Involvement in a structural resistance training program 6 months prior to the start of the experimental trial
* Any kind of injury/incapability that is a contra-indication to perform high-intensity resistance exercise
* Intake of any performance enhancing medication or nutritional supplement 6 months prior to the start of the experimental trial
* Use of PEA supplements or CBD related products (including CBD oil, cannabis or other substances containing cannabinoids) 1 year prior to the start of the experimental trial
* Blood donation within 3 months prior to the start of the experimental trial

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Isometric muscle strength | 4 months
  Maximal isometric peak torque (N x m) assessed via Promett
Eccentric muscle strength | 4 months
  Eccentric isometric peak torque (N x m) assessed via Promett
Concentric muscle strength | 4 months
  Concentricisometric peak torque (N x m) assessed via Promett
Jump height | 4 months
  2 leg jump height on a force platform (m)
Plasma concentrations of PEA, creatine kinase (CK), IL-6 and TNFα | 4 months
  Plasma concentrations of PEA, creatine kinase (CK), IL-6 and TNFα
Muscle inflammatory signaling | 4 months
  pro- and anti-inflammatory cytokine expression (TNFα, IL-6, IL-10, IL-4) assessed via western blotting and PCR (arbitrary units)
Muscle immune cell infiltration | 4 months
  immune cell infiltration (macrophages and neutrophils) (number/area) assessed via histological analyses of muscle biopsies

SECONDARY OUTCOMES:
Dietary behaviour | 4 months
  micro and macronutrient intake will be assessed via an online application in which the participants report all their dietary intake (expressed as (relative) energy (contribution), e.g. kcal)
Perceived sleep quality | 4 months
  Sleep quality will be assessed via a questionnaire (arbitrary units)
Perceived sleep quantity | 4 months
  Sleep quantity will be assessed via a questionnaire (hours/night)

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Koppo, PhD, Principal Investigator — KU Leuven
Locations (1):
- Exercise Physiology Research Group, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No